CLINICAL TRIAL: NCT05554328
Title: A Randomized Trial of Selumetinib and Olaparib or Selumetinib Alone in Patients With Recurrent or Persistent RAS Pathway Mutant Ovarian and Endometrial Cancers: A ComboMATCH Treatment Trial
Brief Title: Testing the Use of the Combination of Selumetinib and Olaparib or Selumetinib Alone Targeted Treatment for RAS Pathway Mutant Recurrent or Persistent Ovarian and Endometrial Cancers, A ComboMATCH Treatment Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-06841; NCI-2022-06841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-N4 (Other: NRG Oncology); EAY191-N4 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (selumetinib, olaparib) (Experimental): Patients receive selumetinib PO BID and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Drug: Selumetinib Sulfate
- Arm II (selumetinib) (Active Comparator): Patients receive selumetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may elect to cross over to Arm I provided they have not had dose limiting toxicities to monotherapy selumetinib. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Selumetinib Sulfate

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration or biopsy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm I (selumetinib, olaparib)
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate

SUMMARY:
This phase II ComboMATCH treatment trial compares selumetinib plus olaparib to selumetinib alone in women with endometrial or ovarian (fallopian tube and primary peritoneal) cancer that has come back (recurrent) or that remains despite treatment (persistent) and harbors a mutation in the RAS pathway. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Olaparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. The addition of olaparib to selumetinib could increase the percentage of tumors that shrink as well as lengthen the time that the tumors remain stable (without progression) as compared to selumetinib alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare progression free survival of combination of olaparib and selumetinib sulfate (selumetinib) to selumetinib alone in patients with RAS mutant ovarian cancer. (Cohort 1) II. Compare progression free survival of combination of olaparib and selumetinib to selumetinib alone in patients with RAS mutant endometrial cancer. (Cohort 2)

SECONDARY OBJECTIVES:

I. Determine safety of both arms per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

II. Compare objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between the two arms.

III. Determine rate of objective response per RECIST 1.1 in those patients that crossover from the single agent arm to the combination arm.

IV. Report duration of response of the two treatment arms. V. Collect tissue and provide it to the ComboMATCH Registration protocol to assess concordance between the diagnostic tumor mutation profile generated by the designated laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor (ct)DNA mutation profile from plasma, as described in ComboMATCH Registration protocol. For this treatment substudy, the outcome objective will be to report the proportion of cases providing sufficient tissue for that integrated scientific activity in the ComboMATCH Registration protocol.

TRANSLATIONAL OBJECTIVE:

I. To assess association of baseline genomic and transcriptomic status with response and resistance to therapy.

OUTLINE: Patients in both cohorts are randomized to 1 of 2 arms.

ARM I: Patients receive selumetinib orally (PO) twice daily (BID) and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as echocardiogram (ECHO) or multigated acquisition (MUGA), and computed tomography (CT) scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.

ARM II: Patients receive selumetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may elect to cross over to Arm I provided they have not had dose limiting toxicities to monotherapy selumetinib. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-N4 based on the presence of an actionable mutation as defined in EAY191
* Patients must be enrolled on the ComboMATCH Master Registration Trial EAY191
* Patients must have RAS pathway mutations as determined by the ComboMATCH screening assessment

  * Cohort 1: Patients with histologically confirmed RAS pathway mutant ovarian, primary peritoneal, or fallopian tube ("ovarian") cancer (activating mutations in KRAS, NRAS, HRAS, BRAF, MEK1, MEK2, or inactivating mutations in NF1)
  * Cohort 2: Patients with histologically confirmed RAS pathway mutant endometrial cancer (activating mutations in KRAS, NRAS, HRAS, BRAF, MEK1, MEK2, or inactivating mutations in NF1)
* Patients must have disease that can be safely biopsied and agree to a pre-treatment biopsy or, if disease cannot be safely biopsied, have archival tissue available from within 12 months prior to the date of registration on the ComboMATCH Registration Trial (EAY191)
* Patients must have progressed after first-line treatment for recurrent or persistent disease
* Patients with ovarian cancer should not be eligible for further platinum-based therapy
* Patients with endometrial cancer must have received or been offered an immune oncology agent (alone or in combination with lenvatinib) unless there are existing contraindications for immune oncology agents or lenvatinib
* Patients may have received unlimited prior therapy
* Patients must have measurable and biopsiable disease. Measurable disease is defined by RECIST 1.1 as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be > 10 mm when measured by CT, magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or > 20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI

  * Patients must have at least one "target lesion" separate from the lesion to be biopsied to be used to assess response on this protocol as defined by RECIST version 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Prior therapy must have been completed at least four weeks prior to registration
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* Hemoglobin (Hgb) >= 9.5 g/dL with no blood transfusion in the past 28 days (within 14 days prior to registration)
* Platelets >= 100,000/mcl (within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to registration)
* Patients must have creatinine clearance estimated of >= 50 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test (within 14 days prior to registration)
* Total bilirubin level =< 1.5 x institutional upper limit of normal (ULN) or =< 3 x ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (within 14 days prior to registration)
* Patients must be able to swallow and retain oral medications and be without gastrointestinal illnesses that would preclude absorption of selumetinib or olaparib
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Women of childbearing potential (WOCBP) must agree to use two forms of birth control (hormonal or barrier method of birth control; abstinence) during the study and for 6 months after completing treatment

  * Non-sterilized male partners of WOCBP (including males sterilized by a method other than bilateral orchidectomy e.g., vasectomy) who intend to be sexually active with a female partner must be using an acceptable method of contraception such as male condom plus spermicide (condom alone in countries where spermicides are not approved) from the time of screening throughout the total duration of the study and the drug washout period (at least 6 months after the last dose of study intervention) to prevent pregnancy in a partner. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Vasectomized (i.e., sterile) males are considered fertile and should still use a male condom plus spermicide as indicated above during the clinical study
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated

  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required during the first cycle of therapy

  * Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression
  * Extra caution should be taken with olaparib, as it crosses the blood brain barrier and can cause edema in brain metastases
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have received any MEK inhibitors
* Patients who have progressed while receiving a PARP inhibitor
* Patients who have received chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to registration
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients with uncontrolled intercurrent illness
* Patients with >= grade 2 neuropathy within 14 days of registration
* Patients with severe (Child-Pugh C) liver dysfunction
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib and selumetinib or any excipients thereof
* Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents

  * Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to study enrollment even if less than 100% of the daily recommended dosing for vitamin E
  * Vitamin E must not be taken in the 7 days prior to initiation of treatment with selumetinib
* Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or known moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, Fluconazole, verapamil). The required washout period prior to starting olaparib is at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication
* Concomitant use of strong CYP2C19 inhibitors (e.g., ticlopidine) or moderate CYP2C19 inhibitors (e.g., omeprazole). The required washout period prior to starting selumetinib is at least 14 days or 5 half-lives (whichever is longer) before the first dose of study medication
* Have received or are receiving an investigational medicinal product (IMP) or other systemic anti-cancer treatment (including chemotherapy, immunotherapy, targeted therapy, biologic therapy, tumor embolization, or monoclonal antibodies) within 4 weeks prior to registration, or within a period during which the IMP or systemic target treatment has not been cleared from the body (e.g., a period of 5 'half-lives'), whichever is longer
* Known myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Patients who have had previous organ transplant, allogenic bone marrow transplant or double umbilical cord blood transplantation
* Patients who have had whole blood transfusion within 28 days prior to registration
* Patients with ophthalmological conditions as follows:

  * Current or past history of retinal pigment epithelial detachment/central serous retinopathy or retinal vein occlusion.
  * Intraocular pressure > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of intraocular pressure [IOP]). Subjects with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the study chair
  * Patients with any other significant abnormality on ophthalmic examination should be discussed with the study chair for potential eligibility
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or longstanding orbito-temporal plexiform neurofibroma (PN) (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Patients with severe, active co-morbidity defined as any of the following:

  * History and/or confirmed pneumonitis
  * Uncontrolled hypertension (blood pressure [BP] >= 150/90 mmHg despite medical therapy)
  * Acute coronary syndrome within 6 months prior to registration
  * Uncontrolled atrial fibrillation
  * Known family history of long QT syndrome
* Women who are pregnant or unwilling to discontinue nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | The duration of time from enrollment to the date of progression or death, whichever occurs first, assessed up to 5 years
  Disease progression will be defined using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria, as determined by the treating physician. The primary analyses will be based on logrank tests stratified by the stratification factors as recorded at randomization. All enrolled patients will be included, regardless of compliance with their assigned study regimen. Patients will be grouped by their randomized treatment for intention-to-treat analyses. Treatment hazard ratios and 90% confidence intervals will be estimated using proportional hazards models specified with a main-effect for the randomized treatment assignment (experimental versus [vs] reference), and stratified using the stratification factors recorded at randomization. Treatment group differences will be graphed using Kaplan-Meier methods.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | Up to 5 years
  The safety population will support these analyses. The nature, frequency, and degree of toxicity will be tabulated at the System Organ Class and AE-specific term levels using Common Terminology Criteria for Adverse Events v5.0. Each patient will be represented according to the maximum grade observed for each term. Tabulations will show the number and percentage of patients by maximum grade, within the treatment group received, regardless of the randomized treatment assignment.
Objective response rate (ORR) between two arms | Within 6 months of the date of last enrollment
  ORR is defined as the binomial proportion of evaluable patients with a best overall response of complete response (CR) or partial response (PR) (by RECIST 1.1) within 6 months of the date of the last enrollment. Responses reported by the treating physician will be used for these analyses. The ORR estimates by treatment arm will be supported by their 2-sided, 95% Wilson-Score confidence intervals. The relative odds of response in the experimental arm (vs the reference arm) will be estimated using a multivariable logistic regression model specified with main effects for the randomized treatment assignment and covariate adjustments for the stratification factors reported at baseline.
ORR in crossover patients | Up to 5 years
  Determined by RECIST 1.1. The crossover population will support these analyses. The same evaluation criteria for ORR in the measurable disease population will be applied to the crossover population. These analyses will be done separately for each cohort.
Duration of response of both arms | The time from documentation of either PR or CR until disease progression or death, whichever is observed first, assessed up to 5 years
  These analyses will be supported by patients in the measurable disease population who have a best overall response of PR or CR. Treatment group differences in response duration will be graphed using Kaplan-Meier methods and compared using logrank tests, stratified by the stratification factors defined at randomization. The relative hazards of progression or death in the experimental group (vs the reference group) will be estimated using a multivariable proportional hazards regression model specified with main effects for the treatment indicators and covariate adjustments for the stratification factors reported at baseline. These analyses will be done separately for each cohort.

OTHER OUTCOMES:
ORR | Up to 5 years
  Defined as the binomial proportion of patients with a best overall response of CR or PR. Defined using RECIST 1.1 criteria. Roughly 10 genomic and transcriptomic measures are expected to present as dichotomous factors. When 3 or more levels are presented, the relatively small sample sizes will likely require collapsing down to 2 levels. If presented as continuous variables, the median of the observed values will classify evaluable patients as having wild-type (WT) or mutated expression.
Resistance to therapy | Up to 5 years
  Defined as the proportion of patients with best overall response of disease progression. Defined using RECIST 1.1 criteria. Roughly 10 genomic and transcriptomic measures are expected to present as dichotomous factors. When 3 or more levels are presented, the relatively small sample sizes will likely require collapsing down to 2 levels. If presented as continuous variables, the median of the observed values will classify evaluable patients as having WT or mutated expression.
Concordance between the diagnostic tumor mutation profile, biopsy mutations, and pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutations | Up to 5 years
  Assess the concordance of the diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment ctDNA mutation profile.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — NRG Oncology
Locations (296):
- United States (294):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Tufts Medical Center Cancer Center Stoneham, Stoneham, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Memorial Hospital, Marysville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Puerto Rico (2):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Centro Comprensivo de Cancer de UPR, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm